CLINICAL TRIAL: NCT05308966
Title: Multicenter Observational Retrospective French Study in Patients With Previously Untreated, Unresectable Malignant Pleural Mesothelioma Treated With Nivolumab and Ipilimumab Via an Early Access Program
Brief Title: Observational Study in Patients With Previously Unresectable Malignant Pleural Mesothelioma Treated With Nivolumab and Ipilimumab (MESO-IMMUNE)
Acronym: MESO-IMMUNE
Status: Completed | Type: Observational
Sponsor: Groupe Francais De Pneumo-Cancerologie (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: GFPC 04-2021
Record Dates: First submitted 2022-01-17; First posted 2022-04-04 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-08

CONDITIONS: Malignant Pleural Mesothelioma; Unresectable Malignant Neoplasm
Keywords: Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant; Mesothelioma | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient presenting MPS treated with nivolumab and ipilimumab: Adult patients with previously untreated and unresectable Malignant Pleural Mesothelioma (MPM) treated with combination of Nivolumab and Ipilimumab in the setting of the early access program not opposed to the collection of their data
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Observational study without intervention except retrospective and prospective data collection : Patient characteristics, MPM characteristics, Treatment characteristics, Disease progression, Rebiopsy, Post treatments, Adverse events, Date and cause of death, Date of last news ; recorded in electronic case-report forms (eCRF).

SUMMARY:
Meso-Immune is a retrospective study to assess the efficacy and safety of the combination of Nivolumab and Ipilimumab used in first-line treatment of adult patients with unresectable Malignant Pleural Mesothelioma (MPM). This combination of treatments has been approved in Europe since June 2021 based on the results of the CheckMate 743 study. In France, the combination is not yet reimbursed for this population of patients. However, since April 01, 2021, newly diagnosed unresectable MPM patients may be treated with this combination via an early access program.

Meso-Immune study targets these patients included in the early access program with the objective to provide additional results to the CheckMate 743 study and confirm the benefit of using this combination in first-line of treatment in this category of patients.

Total study duration will cover 48 months with an inclusion period of 12 months and a follow-up until 3 years. Patients will be recruited retrospectively starting April 01, 2021 until April 01, 2022.

Meso-Immune study will be proposed to all the GFPC centers that have already included patients in the early access program and other centers wishing to participate, in order to analyze a minimum of 150 patients. The total number of sites is evaluated at around 120.

The principal investigator in each center will identify the patients eligible for the Meso-Immune study and will inform them on the study according to the local regulations.

Patient follow-up will be pursued regularly, in in-patient and out-patient clinics, according to the usual practices of the physicians in each participating center. Reevaluation workups will be pursued according to the practices of each center.

The information related to Patient characteristics, MPM characteristics, Treatment characteristics, Disease progression, Rebiopsy, Post treatments, Adverse events, Date and cause of death, Date of last news will be recorded in electronic case-report forms (eCRF).

Qualitative variables will be presented descriptively in the principal analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patient with previously untreated and unresectable Malignant Pleural Mesothelioma treated with combination Nivolumab and Ipilimumab in the setting of the early access program
* Patient enrolled in the French National Health Insurance program or with a third-party payer
* Patient not opposed to the collection of his/her data (an information sheet will be to all living patients; for those who died, documented opposition to data collection in his/her medical file is not required)

Exclusion Criteria:

* Patient under curatorship or guardianship
* Patient's explicit refusal to collect his / her data
* Patients not managed at the investigating center and not followed by a center investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with previously untreated and unresectable Malignant Pleural Mesothelioma treated with combination Nivolumab and Ipilimumab in the setting of the early access program not opposed to the collection of his/her data
Sampling Method: Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2025-08-27 (Actual); Study Completion 2025-08-27 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival assessed locally | time from first dose of combination Nivolumab-Ipilimumab to first documentation of disease progression or to death from any cause evaluated through the total duration of the study (up to 48 months)
  Progression free survival as assessed by the investigator, defined as the time from first dose of combination Nivolumab-Ipilimumab to first documentation of disease progression or to death from any cause, whichever came first

SECONDARY OUTCOMES:
Potential professional exposure(s) | At Baseline
  Unresectable Malignant Pleural Mesothelioma Patients' characteristics based on data collected from the patient medical notes. Qualitative parameters will be expressed as numbers, percentages and 95% confidence intervals.
Eastern Cooperative Oncology Group performance status (PS) | At Baseline
  Unresectable Malignant Pleural Mesothelioma Patients' characteristics based on data collected from the patient medical notes. Quantitative parameters will be expressed as means, standard deviations or medians and interquartile ranges.
Body weight | At Baseline
  Unresectable Malignant Pleural Mesothelioma Patients' characteristics based on data collected from the patient medical notes expressed in kilograms. Quantitative parameters will be expressed as means, standard deviations or medians and interquartile ranges.
Body mass index (BMI) | At Baseline
  Unresectable Malignant Pleural Mesothelioma Patients' characteristics based on data collected from the patient medical notes. The BMI is defined as the body mass divided by the square of the body height, and is expressed in units of kg/m 2, resulting from mass in kilograms and height in metres. Quantitative parameters will be expressed as means, standard deviations or medians and interquartile ranges.
Smoking status | At Baseline
  Unresectable Malignant Pleural Mesothelioma Patients' characteristics based on data collected from the patient medical notes. Qualitative parameters will be expressed as numbers, percentages and 95% confidence intervals.
Medical history | At Baseline
  Unresectable Malignant Pleural Mesothelioma Patients' characteristics based on data collected from the patient medical notes. Qualitative parameters will be expressed as numbers, percentages and 95% confidence intervals.
Comorbidities | At Baseline
  Unresectable Malignant Pleural Mesothelioma Patients' characteristics based on data collected from the patient medical notes. Qualitative parameters will be expressed as numbers, percentages and 95% confidence intervals.
Past history of cancer or auto-immune disease | At Baseline
  Unresectable Malignant Pleural Mesothelioma Patients' characteristics based on data collected from the patient medical notes. Qualitative parameters will be expressed as numbers, percentages and 95% confidence intervals.
Overall Survival (OS) | From first dose of combination Nivolumab-Ipilimumab to the end of the study (up to 48 months)
  OS defined as the time from first treatment start to death for any cause expressed in months
Objective Response Rate (ORR) | From first dose of combination Nivolumab-Ipilimumab to the end of the study (up to 48 months)
  Objective Response Rate (ORR): best overall response of complete response (CR) or partial response (PR) to a first line of treatment using i-RECIST criteria as assessed locally
Safety of combination Nivolumab-Ipilimumab | From first dose of combination Nivolumab-Ipilimumab up to 100 days after the last treatment dose administration, up to 48 months (study duration)
  Data on adverse events (AEs) will be collected, and relatedness of these events to the use of drugs associated with this study (where applicable) will be assessed.
Treatment duration | From first dose of combination Nivolumab-Ipilimumab to the end of treatment, up to 48 months (study duration)
  Time to treatment failure, defined as the time from the first dose of combination Nivolumab-Ipilimumab to disease progression locally assessed, death, non-objection withdrawn, adverse event, lost to follow-up or initiation of another anticancer treatment.
Reasons for treatment discontinuation | From first dose of combination Nivolumab-Ipilimumab to the end of treatment, up to 48 months (study duration)
  Reasons for treatment discontinuation will be collected and recorded in the e-CRF
Post-progression treatments | From first dose of combination Nivolumab-Ipilimumab to the end of the study (up to 48 months)
  The name, start and end date, of treatments initiated after the disease progression of the patient will be collected and recorded in the e-CRF. Date of progression for these treatments will be reported as well.
Treatment outcome in terms of PFS in subgroups of patients according to patient's characteristics: elderly patients (age >80 years old), patients with performance status >1, patients with comorbidities | From first dose of combination Nivolumab-Ipilimumab to the end of the study (up to 48 months)
  Treatment outcome in terms of progression free survival as assessed by the investigator, defined as the time from first dose of combination Nivolumab-Ipilimumab to first documentation of disease progression or to death from any cause, whichever came first
Treatment outcomes in terms of AEs in subgroups of patients according to patient's characteristics: elderly patients (age >80 years old), patients with performance status >1, patients with comorbidities | From first dose of combination Nivolumab-Ipilimumab to the end of the study (up to 48 months)
  Treatment outcome in terms of proportion (%) of patients with any adverse event (AE) and number and severity of events per subgroup of patients

CONTACTS AND LOCATIONS:
Overall Officials: Christos CHOUAID, Study Chair — Groupe Français de Pneumo-Cancérologie (GFPC)
Locations (63):
- France (63):
  - CHU du Pays d'Aix, Aix-en-Provence
  - CH Albi, Albi
  - CHU Angers, Angers
  - CH Argenteuil, Argenteuil
  - CH Avignon, Avignon
  - CH Bastia, Bastia
  - CH Bayonne, Bayonne
  - CHU Besançon, Besançon
  - Clinique Ambroise Paré, Beuvry
  - CH Bligny, Bligny
  - Clinique Bordeaux, Bordeaux
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - CHU Morvan, Brest
  - Clinique Pasteur, Brest
  - Hôpital Louis Pradel, Bron
  - CHU Caen, Caen
  - CH Cannes, Cannes
  - CH du Cotentin, Cherbourg
  - CHU Hôpital Montpied, Clermont-Ferrand
  - Unicancer, Clermont-Ferrand
  - Hôpital Louis Pasteur, Colmar
  - CH Dijon Bourgogne, Dijon
  - CH Eure-Seine, Évreux
  - Clinique Gentilly, Gentilly
  - CHD les Oudaries, La Roche-sur-Yon
  - GH Le Havre, Le Havre
  - CH du Mans, Le Mans
  - CH Libourne, Libourne
  - CHU Lille, Lille
  - CH de Longjumeau, Longjumeau
  - Hôpital du Scorff, Lorient
  - Centre Léon Bérard, Lyon
  - IPC, Marseille
  - Hôpital Nord, Marseille
  - CAC Mougins, Mougins
  - CH Nevers, Nevers
  - Clinique Saint Georges, Nice
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Hôpital Cochin, Paris
  - Hôpital Bichat, Paris
  - Hôpital La Pitié-Salpêtrière, Paris
  - GH Paris Site St Joseph, Paris
  - Hôpital Haut-Lévèque - Groupe Hospitalier SUD, Pessac
  - CHU La Mileterie, Poitiers
  - CH Annecy Genevois, Pringy
  - CH Cornouaille, Quimper
  - CHU Ponchailloux, Rennes
  - Clinique Saint Grégoire, Rennes
  - Hôpital Charles Nicolle, Rouen
  - Hôpital privé de la Loire, Saint-Etienne
  - Insititut de Cancerologie de l'Ouest, Saint-Herblain
  - HIA Begin, Saint-Mandé
  - Clinique de l'Estuaire, Saint-Nazaire
  - CH St Quentin, Saint-Quentin
  - CH de Saint Malo, St-Malo
  - Les Hôpitaux Universitaires de Strasbourg, Strasbourg
  - CHITS Toulon Sainte Musse, Toulon
  - HIA St Anne, Toulon
  - Hôpital Larrey, Toulouse
  - CHRU Bretonneau, Tours
  - CH Villefranche, Villefranche-sur-Saône
  - CH Villeurbanne, Villeurbanne

IPD SHARING:
Plan to Share IPD: No